CLINICAL TRIAL: NCT05196893
Title: Link for Schools: A System to Prevent Violence and Its Adverse Impacts
Brief Title: Link for Schools: an Evaluation of a Tiered Staff Training Program and Student Intervention to Prevent Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Heimer (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency); University of Minnesota (Other); Cedar Rapids Community School District (Unknown)
Responsible Party: Sponsor-Investigator, Karen Heimer, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201705712; 2016-CK-BX-0006 (Other Grant/Funding Number: National Institute of Justice)
Record Dates: First submitted 2021-12-07; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Risk Reduction Behavior
Keywords: School violence prevention
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: This study is a two-level randomized intervention trial of students from 12 schools in three clusters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Student Intervention Group (Experimental): Eligible students who were randomized into an immediate intervention group, and received intervention from school staff who received specialized intervention training starting in the fall semester of the academic year. Students from two clusters of schools received staggered intervention (Cluster 1 starting in year 1, and Cluster 2 starting in year 2). School staff recorded details of intervention sessions in a case management tool, and administrative records were maintained by the school district, for evaluation purposes.
  Interventions: Behavioral: Link Intervention
- Wait-list Student Intervention Group (Experimental): Eligible students who were randomized into a wait-list intervention group, and received intervention from school staff who received specialized intervention training starting in the spring semester of the academic year. Students from two clusters of schools received staggered intervention (Cluster 1 starting in year 1, and Cluster 2 starting in year 2). School staff recorded details of intervention sessions in a case management tool, and administrative records were maintained by the school district, for evaluation purposes.
  Interventions: Behavioral: Link Intervention
- Within School Student Control Group (No Intervention): Eligible students who were randomized into either the immediate or wait-list intervention groups, but did not receive intervention from school staff. This was used as a control group instead of an intended 3rd Cluster, which ultimately was not a comparable control based on enrollment and demographic characteristics.

INTERVENTIONS:
Behavioral: Link Intervention — Eligible students met with staff trained in specialize intervention skills. Staff met with students multiple times per month, for approximately 10-30 minutes. During these sessions, staff had conversations with students, using intervention communication skills, assessed student stress, and implemented strategies for behavior change. Details of the sessions were recorded in a case management tool. Students were referred to additional resources, as necessary, and these referrals were also recorded. Rates of student office referrals were assessed over time.
  Arms: Immediate Student Intervention Group; Wait-list Student Intervention Group

SUMMARY:
The University of Iowa in collaboration with the Cedar Rapids Community School District (CRCSD) conducted an effectiveness study to test a theory-based system, called Link, that trained school staff to provide a sustainable infrastructure of support for youth at-risk of violence. Our purpose was to prevent and intervene in violence that impacts students, and to adopt cost-effective school-based violence prevention strategies.

The research team conducted a randomized intervention trial with three "clusters" of within the CRCSD using the procedures described in the following paragraph. Each cluster consisted of a middle school and three "feeder" elementary schools. Implementation of the program began in Fall 2017 at Cluster 1, Fall 2018 at Cluster 2, and Cluster 3 remained a control site and received no intervention.

Program Implementation, by Cluster:

A series of videos were produced by the University of Iowa team in conjunction with the CRCSD, and were offered as a training opportunity to school staff. The series of video trainings include: Trauma Informed Care (TIC) video to be viewed by all staff; and a Link Program training video for select staff.

TIC video instructions was required of all staff during a workshop session. Participants were invited to complete a post-training evaluation survey following the viewing of the TIC video, for research.

Concurrent with the delivery of the Trauma Informed Care video training, select staff were identified by the CRCSD research team to become Link interventionists, by participating in specialized training of the Link system using the Link Program video and in-person trainings. These interventionists had a dual role as a study participant and as a member of the research team. These interventionists were provided 4 in-person trainings throughout the school year that included training in child assent procedures, and Link Program training. These interventionists were invited to complete pre/post evaluation surveys at each training session, for research.

Targeted Research Intervention:

Following the Link Program Training, the CRCSD research team randomly assigned a case load of students to the Link interventionists with whom they used the Link Program skills. Following each student encounter, the interventionist completed a Link Case Management Tool for process evaluation. Link interventionists were also invited to complete a pre-evaluation survey prior to Link Program training, and post-evaluation surveys following training sessions.

Data collected for the targeted student intervention included: primary data in the form of a Link Case Management Tool completed by a Link interventionist following each student encounter; secondary data in the form of existing school administrative data sources (i.e., enrollment and office referrals).

DETAILED DESCRIPTION:
Program implementation and the targeted student intervention were implemented using a staggered approach.

Cluster 1 began study procedure in 2017, and the process is outlined below.

Program Implementation:

Trauma Informed Care Training: Following consent, staff participants viewed a Trauma Informed Care (TIC) training video (TIC video available for review at: https://publichealth.uicapture.uiowa.edu/Panopto/Pages/Sessions/List.aspx?folderID=e4d017e6-6133-4d0b-819d-495f72c74284) that was delivered at a staff in-service session organized by the school district. All participants were invited to complete an anonymous "TIC post-training evaluation" survey immediately following TIC video viewing; those participating in in-person training will complete a paper survey.The survey took approximately 5-10 minutes to complete.

Specialized Link Interventionist Training- Session 1: Identified Link Interventionists were provided training by UI IRB and the UI Research team, for their role as research team members for purposes of assenting students participants, and to be trained in study protocol. The research team presented a group presentation about the research study, and following consent, participants were invited to complete an anonymous "Link_pre-program evaluation" survey. The survey took approximately 5-10 minutes to complete.

Session 2: The Link Program training session consisted of a combination of Link video training (Link training video available for viewing at: https://publichealth.uicapture.uiowa.edu/Panopto/Pages/Sessions/List.aspx?folderID=e4d017e6-6133-4d0b-819d-495f72c74284) and in-person training conducted by the UI research team. Participants were invited to complete an anonymous "Link_post training evaluation_initial" survey at the end of the session. The survey took approximately 5-10 minutes to complete. This training session lasted approximately 2 hours and occurred during an in-service training session scheduled by the school district. Following this training session, participants were randomly assigned a case load of students with which they used the Link Program skills. Following each student encounter, the interventionist completed a "Link Case Management Tool" for process evaluation. This tool took approximately 5-10 minutes to complete.

Session 3: Approximately 6 weeks following the initial training session, a follow-up training session was conducted. This training session consisted of video training and in-person training. Additional video training consisted of reviewing specific student scenario videos and other additional videos developed by the research team (7 scenarios and "Tools for You" are available for review at: https://publichealth.uicapture.uiowa.edu/Panopto/Pages/Sessions/List.aspx?folderID=e4d017e6-6133-4d0b-819d-495f72c74284). Participants were invited to complete an anonymous "Link_post training evaluation_follow up" survey at the end of the session. The survey took approximately 5-10 minutes to complete. This training session will last approximately 2 hours and occurred during an in-service training session scheduled by the school district.

Session 4: At the end of the school year, a final training session was conducted. This training session consisted of a de-briefing discussion about challenges, successes, and future implementation. Participants were invited to complete an anonymous "Link_post program evaluation" survey at the end of the session. The survey took approximately 5-10 minutes to complete. This training session lasted approximately 1 hour and occurred during an in-service training session scheduled by the school district. Due to school cancellation because of the COVID-19 response, this training session was conducted remotely via zoom during the final year of the study; participants were able to join the training session using a laptop or phone. The research team provided a zoom link to the school district project manager, who emailed a meeting invitation to all program interventionists/participants. Following the training session, a survey link to the evaluation survey was emailed to participants via REDCap's automated survey function and completed electronically. Data was stored in a REDCap database maintained by the University of Iowa.

These Link interventionist training sessions were audio recorded for training content analysis.

Targeted Student Intervention The school district research team maintained a list of students in Clusters 1, 2, and 3 schools whose parents have provided consent for participation, and met eligibility criteria. Students were then assigned to randomization arms by the research team.

Immediate intervention group: Following assent by the Link Interventionist, the student had a conversation with the interventionist in which the interventionist used specific communication skills they learned through their training described above. The interventionist may or may not have used specific tools they were exposed to during the training sessions (stress screener, etc.) and referred the child to additional resources as necessary. The student subject was invited to meet with the interventionist several times (up to 2 times per week) during the remainder of the school year. These encounters were approximately 10-30 minutes in length, and occurred during the school day in a private location determined by the interventionist and the school district research team. The student was referred to additional resources, as necessary, and as a result of the meetings.

Wait-list control: These students were approached for intervention the semester following the implementation of the intervention, and interventionists used the same procedures described for the immediate intervention group. While on the wait-list, students assigned to this intervention arm received the same standard services offered by the school district to students at control group schools. This multi-level wait-list design (both at Cluster and student level) is ideal for evaluating the effectiveness of a program that is realistically rolled out over time. The wait-list also allows for comparisons between students who receive support vs. those who do not, and comparisons of students in a mature program vs. newly implemented program. The wait-list is an ethical approach used in other intervention evaluation studies of mental health treatment programs for at-risk children exposed to violence. Due to school cancellation due to COVID-19 response, interventionists contacted parents via phone (numbers are available to school staff in PowerSchool) to check-in with the family and student. During this phone call, the interventionists assessed whether the student was interested in continuing the intervention electronically (phone or web meeting). Depending on the students' preference, the interventionist then conducted any future session via phone (using the phone number listed in PowerSchool) or web meeting (an email invitation was sent to the student participant's school-based email address from the interventionist).

Cluster 2: Same procedures as Cluster 1, but commencing the following school year

Cluster 3: Control group, did not receive any training or intervention. During registration at the beginning of the school year, parents were provided a letter via PowerSchool/school district website notifying them that the district will be providing de-identified student data to University of Iowa researchers for research purposes. If parents objected, they were instructed to contact a school district official (listed on the letter), and their student's data would be removed from the data set shared with investigators.

For all clusters, the school district research team provided individual-level data (identified with a student ID number only), sorted by intervention arm, about these students to the UI research team for analysis. This data was in the form of administrative student records (i.e., enrollment, office referrals). The UI research team was not provided a key code for these data.

ELIGIBILITY:
Inclusion Criteria:

1. Elementary and middle school students in grades 3- 8 from clusters 1 and 2, who:

1. Have one or more behavioral referrals in the previous academic year, or
2. Have at least 2 of the following indicators in the previous academic year:

   * attended 80% or less of enrolled school days,
   * were in the 90th percentile and above on tardies,
   * had changed schools since the previous year,
   * were not proficient in ELA (tested only in 6th and 7th grade),
   * were in the 10th percentile or below on math performance,
   * were in the 90th percentile or above on health office visits, or
   * scored positive on the district-administered Pediatric Symptom Checklist.

Exclusion Criteria:

* Students unable to proficiently communicate in English

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 863 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in weekly rate of student office referrals (overall) | weekly, up to 3 academic years
  A mean weekly rate of overall disciplinary office referrals was calculated using counts of student disciplinary office referrals received per academic week, for all referral types. To determine the effectiveness of the intervention in reducing the rate of referrals, negative binomial models were fitted using Generalized Estimating Equations (GEEs); the first model focused on the amount of time each student was in the study and the second model determined if there was a dosage effect with the number of intervention sessions received. Each of these models included covariates (sex, race, and grade level) to account for the differences between the students' demographic groups.
Change in weekly rate of student office referrals (physical aggression) | weekly, up to 3 academic years
  A mean weekly rate of physical aggression office referrals was calculated using counts of student office referrals related to physical aggression, received per academic week. To determine the effectiveness of the intervention in reducing the rate of referrals, negative binomial models were fitted using Generalized Estimating Equations (GEEs); the first model focused on the amount of time each student was in the study and the second model determined if there was a dosage effect with the number of intervention sessions received. Each of these models included covariates (sex, race, and grade level) to account for the differences between the students' demographic groups.
Change in student K-6 stress screener score | every two weeks, up to 3 academic years
  Score of individual student stress, measured using the Kessler-6 (K-6) "Six Simple Questions" stress screener. Interventionists were trained to assess student stress on an as needed basis during intervention sessions, and on at least two occasions: 1) at the start of the student's intervention (during first session), and 2) prior to ending or tapering intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Heimer, PhD, Principal Investigator — University of Iowa; Marizen R Ramirez, PhD, MPH, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Cedar Rapids Community School District, Cedar Rapids, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be archived with the National Archive of Criminal Justice Data (NACJD). Datasets archived include: all training evaluation datasets, case management data, a dataset about linkages to student supports, secondary student administrative data, and cost data.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made publicly available upon successful curation by NACJD.
Access Criteria: Data will be publicly available.